CLINICAL TRIAL: NCT03050736
Title: An Open Label Trial of Dianhydrogalactitol (VAL-083) and Radiation Therapy in Treatment of Newly Diagnosed GBM Patients With An Unmethylated Promoter of the Methylguanine-DNA Methyltransferase (MGMT) Gene
Brief Title: Safety Study of VAL-083 and Radiotherapy in Patients With Newly Diagnosed GBM Having Unmethylated MGMT Expression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kintara Therapeutics, Inc. (Industry)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DLM-14-001
Record Dates: First submitted 2017-01-27; First posted 2017-02-13 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Glioma; Glioblastoma; Glioblastoma Multiforme; GBM; Brain Cancer
Keywords: Glioma; Glioblastoma; Glioblastoma multiforme; GBM; brain tumor; brain cancer
MeSH Terms: conditions — Glioma; Glioblastoma; Brain Neoplasms | interventions — Dianhydrogalactitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VAL-083 (Dianhydrogalactitol) (Experimental): VAL-083 given by intravenous infusion with a starting dose of 20 mg/m2 IV. Escalating doses to be administered in sequential dose cohorts.
  Interventions: Drug: VAL-083 (Dianhydrogalactitol)

INTERVENTIONS:
Drug: VAL-083 (Dianhydrogalactitol) — VAL-083 given by intravenous infusion with a starting dose of 20 mg/m2 IV. Escalating doses to be administered in sequential dose cohorts.

SUMMARY:
The purpose of this Phase 2, open-label, single-arm study is to determine the safety and the maximal tolerated dose (MTD) of VAL-083 in combination with a standard of care radiation regimen when used to treat newly diagnosed GBM in patients with unmethylated promoter of the methylguanine-DNA methyltransferase (uMGMT) gene. Pharmacokinetic (PK) properties will be explored and tumor responses to treatment will be evaluated.

DETAILED DESCRIPTION:
Malignant gliomas are the most common primary central nervous system tumors found in adults, with WHO Grade IV malignant glioma (GBM) representing the most aggressive and prevalent sub-type of these tumors having one of the worst 5-year survival rates among all human cancers.

Standard therapy for patients with malignant gliomas has traditionally involved maximal surgical resection/debulking of the primary tumor (if feasible), followed by adjuvant radiotherapy over 6-8 weeks, with or without chemotherapy. The oral alkylating agent temozolomide was found to increase median survival when used in combination with radiotherapy, compared to radiotherapy alone, in patients with newly diagnosed GBM. However, expression of O6-methylguanine methyltransferase (MGMT) in GBM has been linked to poor patient outcome in patients treated with temozolomide.

The study drug, dianhydrogalactitol (VAL 083) is a bi-functional N7 DNA alkylating agent which has demonstrated cytotoxic activity that is independent of chemo-resistance due to expression of MGMT. This makes VAL-083 an ideal candidate to treat patients who are unlikely to respond to temozolomide due to MGMT expression in their GBM. Furthermore, VAL-083 acted as a radio-sensitizer at low (1 - 2.5μM) concentrations in all GBM cultures tested.

VAL-083 has been studied extensively in the United States by the National Cancer Institute. The NCI studies suggested that VAL-083 appeared to have activity in some types of cancer (lung and brain), including GBM; however, further VAL-083 research was not pursued in the US due to an increased focus on targeted biologic therapies during that era. VAL-083 has also been studied in the People's Republic of China, where it is currently approved and marketed for treatment of chronic myeloid leukemia and lung cancer. At present, VAL-083 is being studied in clinical trials in the United States as a third-line treatment option for patients with recurrent GBM following failure of surgery, radiation therapy, temozolomide and bevacizumab. Interim results support safety of VAL-083 in this population; to date, a regimen of 40mg/m2/d x 3 days IV in a 21 day cycle has been confirmed to be safe and well tolerated.

This phase 2, open-label, single arm study will be conducted in a dose-escalation cohort scheme to confirm the optimal dose of VAL-083, when administered concurrently with radiation therapy. Dose escalation will proceed in three sequential cohorts, consisting of patients receiving VAL-083 at 20, 30 and 40 mg/m2/d x 3 every 21 days.

This trial will be conducted in 2 parts. Part 1 will consist of 1) a 42-day induction period, during which patients will receive VAL-083 while undergoing radiation treatment at a dose of 2 Gy per fraction given once daily five days per week (Monday through Friday) over a period of six weeks (for a total dose of 60 Gy), followed by 2) adjuvant maintenance therapy with VAL-083 alone, administered daily x 3 IV every 3 weeks at the same assigned dose, for a maximum of 8 maintenance cycles. Part 2 will comprise an expansion phase, in which VAL-083 will be studied in up to 20 additional subjects. The dose of VAL-083 that will be studied in Part 2 will be determined from Part 1.

Patients will undergo safety assessments including physical examinations, vital signs, hematology, serum chemistry, and urinalysis.

In both parts of the study, a pharmacokinetic study may be conducted at treatment Cycle 1 Day 1, in consenting patients. For patients consenting to CSF collection by lumbar puncture, a CSF sample will be obtained after completion of the Cycle 1, Day 3 VAL-083 infusion. These patients will also have a blood sample taken for VAL-083 plasma level after completion of drug infusion.

Response parameters will be evaluated according to the Response Assessment in NeuroOncology (RANO).

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed histologically proven supratentorial GBM
2. Tumor tissue specimens from the GBM surgery or open biopsy must be available for MGMT gene promoter status analysis and central pathology review.
3. Documented unmethylated MGMT gene promoter status
4. Males or females ≥18< 70 years of age.
5. Interval of ≥2 weeks but ≤7 weeks after surgery or biopsy before first administration of study treatment.
6. Cranial MRI must have been performed within 21 days of study entry and MRI must be used throughout the period of protocol treatment for tumor measurement. If the surgical procedure was a resection, cranial MRI performed within 72 hours of resection is preferred
7. Stable or decreasing dose of steroids for ≥5 days prior to randomization.
8. Karnofsky performance score ≥ 70%
9. Patients must begin treatment with VAL-083 chemotherapy no sooner than 2 weeks and no later than 4 weeks from the diagnostic surgery.
10. ANC ≥1,500/ µl
11. Platelet count ≥ 100,000/µl
12. Hemoglobin ≥ 10 gm/dl
13. AST, ALT < 2.5 times ULN
14. Bilirubin < 2.5 ULN
15. Serum creatinine ≤ 1.5x ULN or creatinine clearance > 50 mL/min (measured or calculated by the Cockcroft-Gault formula) (Cockcroft, 1976) at screening

Exclusion Criteria:

1. Prior chemotherapy within the last 5 years.
2. Prior radiation therapy of the head.
3. Receiving concurrent investigational agents or has received an investigational agent within the past 30 days prior to the first dose of VAL-083.
4. Prior systemic anti-angiogenic therapy.
5. Placement of Gliadel® wafer at surgery.
6. Planned surgery for other diseases (e.g. dental extraction).
7. History of recent peptic ulcer disease (endoscopically proven gastric ulcer, duodenal ulcer, or esophageal ulcer) within 6 months of enrollment.
8. History of malignancy. Subjects with curatively treated cervical carcinoma in situ or basal cell carcinoma of the skin, or subjects who have been free of other malignancies for ≥5 years are eligible for this study.
9. History of coagulation disorder associated with bleeding or recurrent thrombotic events.
10. Clinically manifest myocardial insufficiency (New York Heart Association [NYHA] III, IV) or history of myocardial infarction during the past 6 months; or uncontrolled arterial hypertension.
11. Inability to undergo Gd-MRI.
12. Concurrent illness, including severe infection, which may jeopardize the ability of the subject to receive the procedures outlined in this protocol with reasonable safety.
13. Subject is pregnant (positive serum beta human chorionic gonadotropin [b-HCG] test at screening) or is currently breast-feeding, anticipates becoming pregnant/ impregnating their partner during the study or within 6 months after study participation, or subject does not agree to follow acceptable methods of birth control, such as hormonal contraception, intra-uterine pessar, condoms or sterilization, to avoid conception during the study and for at least 6 months after receiving the last dose of study treatment.
14. Current alcohol dependence or drug abuse.
15. Known hypersensitivity to the study treatment.
16. Legal incapacity or limited legal capacity.
17. Presence of any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
18. Signs and symptoms suggestive of transmissible spongiform encephalopathy, or family members who suffer(ed) from such.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-12-17 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Efficacy evaluation of tumor response in patients, as measured by magnetic resonance imaging | Every 42 days while receiving radiotherapy then every 63 days while remaining on study, from patient randomization until study discontinuation for up to 10 months
  Tumor response assessment via MRI, as long as patient continues to demonstrate response or stable disease and tolerates therapy.

SECONDARY OUTCOMES:
Safety evaluation of VAL-083 in combination with a standard radiation therapy, as determined by incidence of patient adverse events and changes in laboratory results, ECG and vital signs | Every 30 days, from patient randomization through 28 days following last study treatment for up to 10 months
  To confirm the safety and tolerability of VAL-083 in combination with a standard of care radiation regimen. Safety will be assessed through summaries of AEs, changes in laboratory test results, ECGs, and changes in vital signs for all patients who receive any amount of VAL-083.
Ctrough | On Cycle 1 Day 1 pre-dose, and 15, 30, 60, 120, 240 and 360 minutes after study drug administration then Cycle 1 Day 2 pre-dose
  Pre-dose plasma concentration of VAL-083
Cmax | On Cycle 1 Day 1 pre-dose, and 15, 30, 60, 120, 240 and 360 minutes after study drug administration then Cycle 1 Day 2 pre-dose
  Maximum observed plasma concentration of VAL-083
Tmax | On Cycle 1 Day 1 pre-dose, and 15, 30, 60, 120, 240 and 360 minutes after study drug administration then Cycle 1 Day 2 pre-dose
  Time of observed Cmax for VAL-083 in plasma
AUClast | On Cycle 1 Day 1 pre-dose, and 15, 30, 60, 120, 240 and 360 minutes after study drug administration then Cycle 1 Day 2 pre-dose
  Area under the concentration-time curve from pre-dose (time 0) to the time of the last quantifiable concentration of VAL-083 in plasma
AUCinf | On Cycle 1 Day 1 pre-dose, and 15, 30, 60, 120, 240 and 360 minutes after study drug administration then Cycle 1 Day 2 pre-dose
  Area under the concentration-time curve extrapolated to infinity for VAL-083 in plasma
CL/F | On Cycle 1 Day 1 pre-dose, and 15, 30, 60, 120, 240 and 360 minutes after study drug administration then Cycle 1 Day 2 pre-dose
  Total oral body clearance at steady state for VAL-083 in plasma
Mean Residence Time | On Cycle 1 Day 1 pre-dose, and 15, 30, 60, 120, 240 and 360 minutes after study drug administration then Cycle 1 Day 2 pre-dose
  AUMC/AUC for VAL-083 in plasma, where AUMC is Area under the Moment Curve
Vz | On Cycle 1 Day 1 pre-dose, and 15, 30, 60, 120, 240 and 360 minutes after study drug administration then Cycle 1 Day 2 pre-dose
  Volume of distribution during the terminal phase of VAL-083 in plasma
Lambda z | On Cycle 1 Day 1 pre-dose, and 15, 30, 60, 120, 240 and 360 minutes after study drug administration then Cycle 1 Day 2 pre-dose
  Terminal elimination rate constant determined by selection of at least three decreasing data points on the terminal phase of the concentration-time curve for VAL-083 in plasma
T½ | On Cycle 1 Day 1 pre-dose, and 15, 30, 60, 120, 240 and 360 minutes after study drug administration then Cycle 1 Day 2 pre-dose
  Terminal elimination half-life of VAL-083 in plasma
Pharmacokinetic profile and dose-exposure relationship of VAL-083 in Cerebral Spinal Fluid (CSF) | Once after completion of Cycle 1 Day 3 infusion
  VAL-083 levels in CSF will be correlated with VAL-083 levels in plasma drawn at Cycle 1 Day 3.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Zhong-ping, M.D., Ph.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No
The Clinical Study Report for this trial will be prepared and provided to U.S. F.D.A. as required by applicable regulatory requirement(s). The trial investigator will be provided a copy of their patient data captured in the electronic data base for this trial.

REFERENCES:
- [Derived] Guo C, Yang Q, Deng M, Qiu X, Wu S, Du X, Sai K, Dai Z, Chen Z, Zhang J, Lin F, Ke C, Xi S, Hu W, Zhou Z, Li J, Cao X, Liao Y, Lv Y, Brown D, Langlands J, Johnson G, Bacha J, Kwan C, Kanekal S, Schwartz R, Chen Z. VAL-083 is effective in patients with newly-diagnosed MGMT-unmethylated glioblastoma: report of phase II study. Discov Oncol. 2025 Dec 12. doi: 10.1007/s12672-025-04235-y. Online ahead of print. PMID 41385182